#### **INFORMED CONSENT**

### The Impact of Reduced Pain among the Poor

#### Introduction

You are being asked if you would like to take part in a study led by researchers from universities in the United States. The study wants to understand the lives of people like you. This document will give you information about this study, which will be read to you now. Please listen and read carefully, and ask questions about anything that you do not understand before deciding whether or not to participate. We are very happy to answer any questions that you have about your choice to participate.

Translation: அமெரிக்காவில் இருக்கிற பல பல்கலைகழகங்களில் இருந்து வந்துள்ள ஆய்வாளர்களால் நடத்தப்படும் ஆய்வுக்கு பங்கெடுக்க விருப்பம் உள்ளதா என்று கேட்டுக்கொள்ளப்படுகிறீர்கள். இந்த ஆய்வு உங்களை போன்றவர்களின் வாழ்வை புரிந்த கொள்ள நடத்த படுவது ஆகும். இப்பொழுது நான் படிக்கும் இந்த ஆவணம் உங்களுக்கு இந்த ஆய்வை பற்றிய தகவலை கொடுக்கும். நீங்கள் இந்த ஆய்வில் பங்கெடுக்கலாமா இல்லையா என்று முடிவு செய்வதற்கு முன் நான் சொல்லுவதை முழுவதும் கவனமாக கேட்கவும்.நீங்கள் பங்கெடுப்பதை பற்றி எதாவது கேள்வி இருந்தால் நாங்கள் அதற்கு சந்தோஷமாக பதில் அளிக்கிறோம்.

### Voluntary participation and withdrawal

Translation: தன்னார்வ பங்கெடுப்பு மற்றும் விலகுதல்

It is your choice whether to participate in the study or not. If you choose to be in this study, you may leave or quit the study at any time without penalty or consequences of any kind.

Translation: உங்கள் பங்கேற்பும் விலகுதலும் உங்கள் சுய விருப்பத்தை சார்ந்தது. நீங்கள் எப்போது வேண்டுமானாலும் இந்த ஆய்வை விட்டு அபராதம்/பின்விளைவு ஏதும் இன்றி விலகி கொள்ளலாம்.

Purpose of the study

Translation: ஆய்வின் நோக்கம்

## INFORMED CONSENT\_EL

The purpose of this study is to learn about some of the issues and challenges that affect the lives and work of flower stringers.

Translation: இந்த ஆய்வின் நோக்கம் பூ தொடுக்கும் தொழிலாளர்களின் வாழ்க்கையும், பொருளாதாரவிளைவுகளை பாதிக்கும் பிரச்சனைகள் மற்றும் சவால்கள் பற்றி படிப்பதே ஆகும்.

### **Procedures**

Translation: செயல்முறை

If you choose to participate in this study we will ask you to do the following things:

Translation: நீங்கள் இந்த ஆய்வில் பங்கெடுக்க தேர்ந்தெடுத்தால் நாங்கள் உங்களை பின் வரும் காரியங்களை செய்ய கூறுவோம்:

Participate in two sessions at this office. Today is the first session, it will last three hours
during which you will take surveys about your life and work as well as undertake a few of
the short tasks. The second day session will be about seven hours long. We will ask you
to string flowers, complete tasks, and take surveys during this time. Most of the activities
will be done twice, i.e. once in the morning and once again in the afternoon. Also, we will
ask you to do a task in which you quickly put one hand in cold water at two points during
the day.

நீங்கஇரண்டு பகுதிகளுக்கு வரவேண்டியதாக **Translation:** இருக்கும்.இது தான்முதல் பகுதி, இந்த 3 மணி நேரத்துல நாங்க உங்களிடம் உங்க வாழ்க்கை மற்றும் உங்க வேலை பற்றியும் சில கேள்விகள் கேட்போம்.இரண்டாவது நாள் 7 மணி நேரம் இருக்கும். கட்ட, சில விளையாட்டு, சில அதுல உங்கள பூ செய்ய சொல்வோம்.கூடவே சில செயல்பாடுகள் கேள்விகளையும்கேட்போம் அதுல சில செயல்பாடுகள் இரண்டுதடவ செய்ற மாதிரி இருக்கும்.அதாவது காலையில ஒரு மற்றும் மதியம் ஒரு தடவ.கூடவே நாங்க உங்கள ஐஸ் தண்ணல் ஒரு நாளைக்கு இரண்டு தடவ உங்க ஒரு கைய வைக்கவும் கேட்போம்.

In addition, on the second day, some participants will be chosen using a lottery to receive tablets that may or may not reduce pain. If you are selected to receive the tablets, you will be asked to take the tablet here in our office. There is a good chance that you may be

### INFORMED CONSENT\_EL

selected to take the tablets as a part of this study, so it is important that you only join the study if you are willing to take the tablets if the lottery assigns you to receive them.

**Translation:** மேலும் இரண்டாவது நாள்லஒரு சில பங்கேற்பாளர்களுக்கு குலுக்கல் முறையில் மாத்திரைகள் வழங்கப்பட்ட வழங்கப்படும். மாத்திரைகள் வலியை குறைக்கவோ அல்லது குறைக்காமல் இருக்கவோ செய்யலாம். நீங்கள் குலுக்கல் முறையில் தேர்ந்தெடுக்கபட்டால் மாத்திரையை உட்கொள்ளும்படி அலுவலகத்தில் கேட்டுக்கொள்ள இங்கு படுவரீகள். மாத்திரை உங்களுக்கு கிடைக்கும் வாய்ப்பு அதிகம், ஆதலால் உங்களுக்கு குலுக்கல் முறையில் மாத்திரை எடுக்க தேர்வு செய்யபட்டால், மாத்திரை எடுக்க விருப்பம் இருந்தால் மட்டுமே இந்த ஆய்வில் சேருங்கள்

### **Potential Risks and Discomforts**

Translation: அபாயங்கள்மற்றும்உபாதைகள்

There are two potential risks that could arise for you from participating in this study:

Translation: நீங்கள் இந்த ஆய்வில் பங்கெடுப்பத்தின் மூலம் இரண்டு அபாயங்கள் உள்ளன.

1. Risks associated with surveys and tasks: We expect that the risk of taking surveys and participating in the tasks are very small and are similar to the ones in your everyday life. We will ask you to complete a task in which you place your hand in cold water. This may be uncomfortable, but it will not harm you.

Translation: ஆய்வுகள்மற்றும்செயல்பாடுதொடர்புடைய ஆபத்துக்கள் நிங்கள் மேற்கூறிய செயல்பாட்டை செய்வதால் மிகவும் குறைந்த மற்றும் நீங்கள் அன்றாட வாழ்வில் சந்திக்கும் ஆபத்துகள் போன்றவையே நாங்க ஐஸ்தண்ணில கை வைக்கிற மாதிரி ஒரு செயல்பாட்டை செய்ய சொல்வோம், அது கஸ்டமா இருக்கலாம் ஆனா உங்க கைய பாதிக்காது.

2. <u>Risks associated with the tablets</u>: The tablets provided in this study are generally considered safe and are available in India in many shops and pharmacies without a prescription from a doctor.

Translation: <u>மாத்திரை சார்ந்த ஆபத்து</u>/ பின்விளைவுகள்:மாத்திரைகள் அனைத்தும் பாதகாப்பானது என உறுதி செய்யப்பட்டது, மேலும் இவை அனைத்தும் மருந்தகங்களில் மருத்துவரின் குறிப்பின்றி வாங்க கூடியவை.

Studies have shown that these tablets are safer than other common painkillers you may know, such as diclofenac (Diclowin Plus). Most common risks associated with such tablets are kidney damage and gastrointestinal discomfort. However, these primarily occur with high-dose prescription use when you take the tablets for a long time. In contrast, today we will only ask you to take one single tablet.

Translation: மற்ற ஆய்வின் அடிப்படையில் இதன் மாத்திரையின்) செய்யப்பட்டது. ஆய்வின்போது பாதகாப்பு உறுதி கொடுக்கப்படும் மாத்திரைகள் அனைத்தும் மற்ற ഖഖി நிவாரணிகளைdiclofenac (Diclowin Plus) விட பாதுகாப்பானவை.அந்த மாத்திரைகளால் பொதுவாக வரக்கூடிய பின் விளைவுகள் என்ன வென்றால் சிறுநீரக பாதிப்பு மற்றும் இரைப்பை கோளாறுகள். எப்படியானாலும், இந்த பாதிப்பு இந்த மாத்திரைகளால் தொடர்ந்து முதன்மையாக அதிக அளவில் ரொம்ப நாளைக்கு எடுத்தாள் மட்டும் முரண்பாடாக இன்று நாங்கள் உங்களை வரும். மாத்திரை மட்டும் தான் எடுக்க சொல்லி கேட்போம்.

Also, we will ask you questions about your medical history to ensure that you do not have any conditions that make you likely to have any risks from taking the tablet.

Translation: மேலும் மருத்துவ வரலாறு பற்றிய கேள்விகள் கேட்டு உங்களுக்கு மாத்திரை எடுப்பதினால் எந்த ஒரு பின்விளைவு வராத மாதிரி உங்க நிலைய தெரிஞ்ச உறுதிப்படுத்துவோம்.

Finally, taking these tablets also involves other very rare potential side effects, such as chest pain, nausea, stomach pain, or loss of appetite. However, doctors have shown that the frequency of such side effects is very low and the government considers the risks to be low enough to allow the sale of these tablets without a prescription at both shops and pharmacies.

Translation: இறுதியாக, மார்பக வலி, குமட்டல், வயிறு வலி அல்லது பசியின்மை போன்ற சில சாத்தியமான பக்க விளைவுகள் அரிதாக வரலாம். எப்படியானாலும்,மருத்துவர் வந்து இந்த மாத்திரியான பக்கவிளைவுகள் ரொம்ப குறைவுனும்,மற்றும் நம்ப அரசாங்கமே இந்த பாதிப்புகளை குறைவானது என நினைச்சு எல்லா மருந்து

கடைகளிலும் மருந்து சீட்டு இல்லாமலே விற்க அனுமதி வழங்கி இருக்கு

We also have a nurse at the study office throughout the day in case you experience any side effects.

Translation: ஓரு வேலை உங்களுக்கு ஏதாவது பின்விளைவுகள் வந்தால் பாக்குறதுக்கு நம்ம ஆபீஸ் ல நாள் முழுவதும் ஒரு நர்ஸ் இருப்பாங்க..

# Payment for Participation பங்கேற்பும் ஊதியமும்

You will be paid for your time here. The lowest payment is Rs. 150 and the normal payment is about Rs. 250. The payment will take place after you are done completing the surveys.

Translation: நீங்க இங்க செலவிடுற நேரத்துக்கு உங்களுக்கு பணம் தந்திடுவோம். குறைந்த பட்ச வருமானம் Rs.150 மற்றும் பொதுவான வருமானம் rs. 250 வரை இருக்கும். உங்களுடைய அனைத்து கேள்விகள் முடிந்த பின்பு நாளின் முடிவில் உங்களுக்கு தொகை தரப்படும்.

The second day, your payment will be different depending on how well you complete the tasks. The lowest payment is Rs. 400 and the normal payment is about Rs. 550. You will also be given 50% of the flowers you strung to take home with you. You may keep or sell these flowers. They are yours to do what you wish with. You will receive a payment of Rs. 70 as a part of your total compensationif you complete all the activities by the end of the day including debriefing. Payments will take place after you are done participating in the study.

Translation: இரண்டாவது நாள், உங்களுக்கு வழங்கப்படும் தொகையானது , நீங்க எவ்ளோ நல்லா செயல்பாடுகளை செய்யரின்களோ அதபொருத்து மாறுபடும் .குறைந்த பட்சம் Rs. 400, முதல்Rs. 550 வரை வழங்கப்படும் .கூடவே உங்களுக்கு நீங்க கட்டற பூவிலிருந்து 50% பூவை நீங்க உங்க வடீடுக்கு எடுத்துட்டு போகலாம். நீங்க அத வெச்சிக்கலாம் இல்ல அத விக்கலாம். அது உங்களுடையது. உங்க விருப்பம். உங்களுக்கு ருபாய் 70 உங்க மொத்த வருமானத்தின்ஒரு பகுதியாக ஆராய்ச்சியின் முடிவில் உங்களுக்கு வழங்கப்படும்.

As described above, you can leave the study at any time without penalty if you are not able to keep going or do not want to keep going. You will be paid for whatever tasks you have completed up to that point.

மேலே சொன்னபடி உங்களுக்கு **Translation:** விருப்பம் இல்லனாலும்,தொடர்ந்து பன்ன புடிக்கலனாலும் நீக எப்போ வேணாலும் *ஆராய்ச்சியிலிருந்து* எந்த அபராதமும் இந்த *ஒ(1*5 இல்லாம விட்டுவிளகலாம். நீங்க எந்த செயல்பாடு வரைக்கும் முடிச்சிங்களோ அதுவரைக்குமான பணத்தை வாங்களாம்.நாளோட கடைசி நேரத்துல நீங்க எல்லா செயளல்பாடுகளையும்,நேர்காணலையும் சேர்த்து முடிச்சு இருந்தா உங்களுக்கு Rs70 கூடுதலாகவே வழங்கப்படும்.

We will also provide, clean water, and snacks while you are the office today. You will also be given lunch for the second day session.

Translation: உங்களுக்கு சுத்தமான தண்ணரீ மற்றும் நொறுக்கு தீனி இன்னைக்கு ஆபீஸ்ல வழங்கப்படும் இரண்டாவது நாள் உங்களுக்கு மதிய உணவும் வழங்கப்படும்

### **Potential Benefits**

Translation: சாத்தியமான நன்மைகள்

As just described, you will be paid for your time today. And if you are selected to receive the tablet it is possible that it will reduce your pain. However, there are no direct benefits for you beyond that. However, this research may help society by collecting information on some of the things that affect the lives and work of flower stringers, which may provide information to NGOs that would be helpful in designing programs to help individuals like yourself and your community.

Translation: இப்போ நாங்க சொன்ன மாதிரி நீங்க இங்க செலவிடுற நேரத்துக்கு பணம் தருவோம் ஒருவேள நீங்க மாத்திரை எடுக்க தேர்வு செய்ய பட்டிங்கன்னா, அது உங்க வலிய குறைக்கலாம். எப்படி பாத்தாலும் இது தாண்டி வேற எந்த ஒரு நேரடி நன்மைகளும் இல்ல மேலும் பூ கட்டறதுனால உங்க வாழ்க்கையும் வேலையும்,பாதிக்குற மாதிரி இருக்குறவை என்ன வென்று இந்த ஆராய்ச்சி மூலமா தகவல சேமிச்சு தன்னார்வ தொண்டுநிறுவனத்துக்கு தீர்வுக்கான வழிகாட்டும். இது உங்கள போன்ற மக்களுக்கும் சமுதாயத்துக்கும் திட்டங்கள வடிவமைக்க உதவியா இருக்கும்.

# **Confidentiality**

Translation: இரகசியத்தன்மை

Any information that is collected during this study and that can be identify a specific person will remain confidential, meaning only the researchers can see it, and it will only be given to others with your permission or as required by law.

Translation: உங்க கிட்ட இருந்து நாங்க கேக்கும் எந்த ஒரு தகவலும் தனி நபர அடையாளம் காற்ற மாதிரி உள்ள தகவல் எல்லாம் ரகசியமாக தான் இருக்கும். அப்படியே வெளில சொல்லுரமதிரியிருந்தா உங்ககிட்ட கேட்டுட்டுதான் சொல்லுவோம் அது சட்டத்துக்கு தேவையானதாக தான் இருக்கும்.

We will take several steps to make sure that the information you give us, including both the information collected during screening and during your participation in this office, is kept private. To do this we will keep your name apart from the other information you give us.

Translation: உங்களிடம் இருந்து "ஸ்க்ரீனிங்", பங்கேற்பின்போது பெறப்பட்ட தகவலையும் ரகசியமாக வைக்க பல்வேறு நடவடிக்கைகள் எடுப்போம். உங்களிடம் இருந்து பெறப்படும் எந்த தகவலிலும் உங்கள் பெயர் இடம்பெறாது.

We will also make sure to lock the document with your name in the filing cabinet so no one outside of the study may see it. Also, unless you would like us to keep your name on a list so that we can contact you about future studies, we will destroy the list of names of people who were in the study when the study is over.

Translation: உங்கள் பெயர் அடங்கிய ஆவணம் பெட்டகத்தில் வைத்து பாதுகாக்கப்படும்.ஆய்வின் முடிவில் பங்கேற்பாளரின் பெயர்கள் நிரந்தரமாக அழிக்கப்படும். நீங்கள் விரும்பினால் உங்களின் தகவலை தொடர்ந்து பாதுகாப்போம். இது பின் வரும் ஆய்வுக்கு நீங்கள் தகுதி அடைய உதவும். எங்க ஆராய்ச்சி முடிந்த பிறகு பங்கேற்ற மக்களுடைய பெயர முழுமையாக அழிச்சுடுவோம்.

We may keep and give others information about study participants as a group. But we will not provide any information that others can use to identify you to other persons or groups.

Translation: பங்கேற்பாளர்களை ஒரு குழுவாக கருதி தகவலை நாங்கள் வெளியிடலாம். ஆனால் எந்நிலையிலும் தனி நபர் தகவல்கள் வெளியிடப்படமாட்டது.

### **Identification of Investigators**

If you have any questions or concerns about the research, please contact:

Blessy Chalcedony, 044 47600844, No. 19 (2nd floor), Mooker Nallamuthu Street, Parrys Corner, Chennai – 600001

### INFORMED CONSENT\_EL

Frank Schilbach, +1-617-715-2969, MIT Department of Economics, 50 Memorial Drive, Building E52 Room 560, Cambridge, MA 02139, USA

# **Emergency Care and Compensation for Injury**

Translation: அவசரசிகிச்சை மற்றும் காயஇழப்பீடு

If you feel you have suffered an injury, which may include emotional trauma, as a result of participating in this study, please contact the person in charge of the study as soon as possible.

Translation: நீங்கள் இந்த ஆய்வின் விளைவாய் காயமடைந்தாலோ/மனதளவில் பாதிப்பை உணர்ந்தாலோ விரைவில் ஆய்வின்பொறுப்பாளரைதொடர்புகொள்ளவும்.

### **Rights of Research Subjects**

Translation: பங்கேற்பாளரின் உரிமை

You are not giving up any legal claims, rights or remedies because of your participation in this research study. If you feel you have been treated unfairly, or you have questions regarding your rights as a research subject, you may contact the following address:

Translation: இந்த ஆய்வில் பங்கெடுப்பதினால் உங்கள் சட்ட இழப்பீடோ/உரிமையோ/ நிவாரணமோ எதுவும் பாதிக்காது. நீங்கள் நியாயமற்ற முறையில் நடத்தபடுவதாய் உணர்ந்தால் நீங்கள் இந்த முகவரியில் தொடர்பு கொள்ளலாம்.

Chairman of the Committee on the Use of Humans as Experimental Subjects, M.I.T., Room E25-143B, 77 Massachusetts Ave,

Cambridge, MA 02139; USA Phone:+1-617-253-6787 Email: fschilb@mit.edu

Sundara Rajan, Institute of Financial Management and Research #4 Second Floor, Buhari Towers, Moores Rd, Thousand Lights, Chennai, Tamil Nadu 600006

Phone: 044 4010 1308 Email: sundar@ifmr.ac.in

## SIGNATURE OF RESEARCH SUBJECT OR LEGAL REPRESENTATIVE

I understand the procedures described above. My questions have been answered to my satisfaction, and I agree to participate in this study. I have been given a copy of this form.

Translation: நான் மேற்கூறிய செயல்முறைகளை புரிந்துகொண்டேன். என் கேள்விக்கான பதில் திருப்திகரமாக அமைந்தது. என் முழு விருப்பதுடன் பங்கேற்க சம்மதிக்கிறேன். இந்த ஆவணத்தின் நகல் என்னிடம் கொடுக்கப்பட்டுள்ளது.

| கொடுக்கப்பட்டுள்ளது. | |
|---|---|
| Note: If the participant is unable to sign, they may provide a thumbprint instead. | |
| Printed Name of Subject | |
| Signature of Subject | Date [DD/MM/YYYY] |
| SIGNATURE OF IN | IVESTIGATOR |
| In my judgment the subject is voluntarily and know the legal capacity to give informed consent to part | |
| Printed Name of Investigator | |
| <br>Signature of Investigator | <br>Date [DD/MM/YYYY] |